CLINICAL TRIAL: NCT03638674
Title: Evaluation of Agreement Between CT Scan and 3D-DXA Measurements on the Lombar Spine
Acronym: 3D DXA SPINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: DMS Apelem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LOCAL/2016/VB-01
Record Dates: First submitted 2018-08-02; First posted 2018-08-20 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Bone Fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2nd lumbar spine acquisition in same position (Active Comparator): spine and hip STRATOS DR + 2nd lumbar spine acquisition in same position (with template)
  Interventions: Other: DXA + CT
- 2nd lumbar spine acquisition (Active Comparator): spine and hip STRATOS DR + 2nd lumbar spine acquisition (no template)
  Interventions: Other: DXA + CT
- 2nd hip acquisition in same position (Active Comparator): spine and hip STRATOS DR + 2nd hip acquisition in same position (with template)
  Interventions: Other: DXA + CT
- 2nd hip acquisition (Active Comparator): spine and hip STRATOS DR + 2nd hip acquisition (without template)
  Interventions: Other: DXA + CT

INTERVENTIONS:
Other: DXA + CT — Two dual-energy X-ray scans + CT scan

SUMMARY:
Dual-energy X-ray Absorptiometry is frequently used to measure bone mineral density. A new medical device, Box 3D DXA, creates a 3D image using a statistics reconstruction model developed on the femur. This new imaging technique does not require additional irradiation and ought to improve bone measures as well as incorporating densitometric parameters into the diagnosis. This study will test the reconstruction of the 3D image from lombar spine measurements and compare accuracy against measurements made using CT scan.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient has been referred by a doctor for a PET/CT (Positron Emission Tomography-Computed Tomography) scan or a SPECT (Single Photon Emission Computed Tomography) scan in the Nuclear Medicine and Medical Biophysics Department of Nimes hospital or a bone scan including a SPECT/CT (single photon emission computed tomography coupled with a CT scan)

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patients is under judicial protection or state guardianship
* The patient is pregnant or breast feeding
* The subject has a observably serious scoliosis
* Subject has previously had spinal or hip surgery
* Subject weighs more than 200kg and/or is more than 2 meters tall by 5+65cm wide and 70cm diameter
* Patient uses an insulin pump or wears an insulin or morphine tubing or any attenuating equipment affecting the hips or lumbar spine
* Subject has already had an X-ray exam using a contrast product such as barium in the 7 days preceding the visit
* Subject having undergone γ radiation exam in the 15 days preceding the visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 60 anatomical females and 60 anatomical males
Enrollment: 120 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Concordance in lombar spine measurements between box 3D-DXA (index test) and CT scan (reference test) | Day 0
  Lin's concordance coefficient
Concordance in lombar spine measurements between box 3D-DXA (index test) and CT scan (reference test) | Day 0
  Bland Altman plot

SECONDARY OUTCOMES:
Reproducibility of the 3D-DXA Spine algorithm for lombar spine measurements | Day 0
  2 acquisitions under the same conditions. Using root-mean-square coefficient of variation to calculate the Least Significant Change
Robustness of 3D-DXA Spine measurement for lombar spine measurements | Day 0
  2 acquisitions under the same conditions. Using interquartile range as a measure of dispersion of the variable
Concordance in femur measurements between box 3D-DXA (index test) and CT scan (reference test) | Day 0
  Lin's concordance coefficient
Concordance in femur measurements between box 3D-DXA (index test) and CT scan (reference test) | Day 0
  Bland Altman plot
Reproducibility of the 3D-DXA Femur algorithm for femur measurements | Day 0
  2 acquisitions under the same conditions. Using root-mean-square coefficient of variation to calculate the Least Significant Change
Robustness of 3D-DXA Femur measurement for femur measurements | Day 0
  2 acquisitions under the same conditions. Using interquartile range as a measure of dispersion of the variable

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, France